CLINICAL TRIAL: NCT01439126
Title: A 40-Week, Phase 4, Double-Blind, Placebo-Controlled, Multicenter, Randomized-Withdrawal Study to Evaluate the Long-Term Efficacy and Safety of KAPVAY™ (Clonidine Hydrochloride) Extended-Release in Children and Adolescents With ADHD
Brief Title: Efficacy & Safety of KAPVAY™ Extended-Release in Children & Adolescents With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Concordia Pharmaceuticals Inc., Barbados (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHN-KAP-401
Record Dates: First submitted 2011-09-13; First posted 2011-09-22 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects on KAPVAY™ (clonidine hydrochloride) (Active Comparator): Subjects in the KAPVAY™ arm receive their optimal dose of KAPVAY™ for the 26-week randomized-withdrawal period (Period 3)
  Interventions: Drug: clonidine hydrochloride
- Subjects on Placebo (Placebo Comparator): Subjects in placebo arm tapered off optimal dose of KAPVAY™ (ie, Period 2 Maintenance Dose) at weekly intervals in decrements of 0.1 mg/day until reaching dose of 0 mg/day; subjects then receive only placebo for the rest of the study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: clonidine hydrochloride — KAPVAY™ (clonidine hydrochloride) 0.1 mg, 0.2 mg, 0.3 mg, or 0.4 mg from Weeks 11-36
  Other Names: KAPVAY™
  Arms: Subjects on KAPVAY™ (clonidine hydrochloride)
Drug: Placebo — KAPVAY™ (clonidine hydrochloride) 0.1 mg, 0.2 mg, or 0.3 mg at Week 11; KAPVAY™ 0.1 mg, KAPVAY™ 0.2 mg, or placebo at Week 12; KAPVAY™ 0.1 mg or placebo at Week 13; placebo from Weeks 14-36
  Arms: Subjects on Placebo

SUMMARY:
The purpose of this study is to determine the long-term efficacy and safety of KAPVAY™ (clonidine hydrochloride) extended-release in children and adolescents with Attention Deficit Hyperactivity Disorder (ADHD)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 6 to 17 years inclusive
* Subject as well as parent/guardian is able to sign the informed assent or consent form
* Subject meets Diagnostic and Statistical Manual of Mental Disorders 4th edition, Text Revision (DSM-IV-TR) criteria for a primary diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), combined subtype, hyperactive/impulsive subtype, or inattentive sub-type based on a detailed psychiatric evaluation using the Shorter version of the Kiddie-Schedule for Affective Disorders and Schizophrenia-Present and Lifetime (MINI-Kid) or DSM-IV TR based checklist for ADHD
* Subject has a minimum of Attention Deficit Hyperactivity Disorder-Rating Scale-4th edition (clinician version) total score of 28 at baseline (Visit 2)
* Subject has a minimum of Clinical Global Impressions-Severity of Illness Scale of 4 at baseline (Visit 2)
* Subject is able to swallow intact tablets based upon interview and screening procedures
* Subject is functioning at an age-appropriate level intellectually with an estimated intelligence quotient of at least 70 based on interview and history
* Subject and parent/guardian understand, are willing, to fully comply with the study requirements, procedures, and restrictions defined in this protocol
* Subject has a supine and standing blood pressure measurement within the 95th percentile for age, gender, and height
* If a female has experienced menarche, she must have a negative serum beta human chorionic gonadotropin pregnancy test at screening (Visit 1), negative urine pregnancy test at baseline (Visit 2), agree to be abstinent from sexual activity that could result in pregnancy, or use acceptable contraceptives throughout the period of the study drug exposure and for 30 days after the last dose of the study drug

Exclusion Criteria:

* Subject has a current comorbid psychiatric condition (except oppositional defiant disorder) that is controlled (requiring a prohibited medication or behavioral modification program) or uncontrolled.
* Subject has any condition or illness including clinically significant abnormal screening (Visit 1) laboratory values that, in the opinion of the investigator, represents an inappropriate risk to the subject and/or could confound the interpretation of the study
* Subject has a known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (eg, clinically significant heart block), exercise-related cardiac events including syncope and presyncope, or clinically significant bradycardia
* Subject is pregnant or nursing (lactating) or deemed by the investigator and staff to be at a significant risk of becoming pregnant.
* Subject has orthostatic hypotension or a known history of controlled or uncontrolled hypertension
* Subject has clinically significant electrocardiogram (ECG) findings as judged by the investigator with consideration of the central ECG laboratory's interpretation.
* Current use of any prohibited medication or other medications including herbal supplements that affect blood pressure, or heart rate, or that have central nervous system effects, or affect cognitive performance such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted); or a history of chronic use of sedating medications (ie, antihistamines) in violation of the protocol specified washout criteria at baseline (Visit 2)
* Subject has used an investigational product within 30 days prior to baseline (Visit 2)
* Subject is significantly overweight based on body mass Index (BMI) for age-and gender-specific charts compiled by Center for Disease Control and Prevention. Significantly overweight is defined as a BMI of ≥95th percentile
* Subject is significantly underweight based on BMI for age-and gender-specific charts compiled by Center for Disease Control and Prevention.
* Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to clonidine hydrochloride
* Clinically important abnormality on drug and alcohol screening (excluding the subject's current ADHD stimulant if applicable) at screening (Visit 1)
* Subject has a history of alcohol, other substance abuse, or dependence as defined by DSM-IV-TR (with the exception of nicotine) within the last 6 months.
* Subject is currently considered a suicidal risk in the opinion of the investigator, has previously made a suicide attempt, has a prior history of, or is currently demonstrating active suicidal ideation based on the Columbia Suicide Severity Rating Scale (C-SSRS).
* Subject has a history of failure to respond to an adequate trial of an alpha 2-agonist with stimulant or non-stimulant drug alone or in combination for the treatment of ADHD.
* Subject has a history of a seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years) or the presence of a serious tic disorder (including Tourette syndrome)
* Subjects who have been treated with an immediate release clonidine and/ KAPVAY™ or guanfacine (INTUNIV™) within the past 30 days

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 34 sites in the US. First patient was enrolled on September 8, 2011 and last patient completed on October 29, 2012
Pre-assignment Details: The study population included male or female subjects 6 to 17 years of age, who met the Diagnostic and Statistical Manual of Mental Disorders 4th Edition Text Revision (DSM-IV-TR) criteria for Attention Deficit Hyperactivity Disorder (ADHD).
Groups:
- Subjects on KAPVAY (Clonidine Hydrochloride): Subjects in the KAPVAY arm received their optimal dose of KAPVAY (as determined after a 4-week, open-label, dose optimization period) for the duration of the 26-week randomized-withdrawal period.
  All subjects were given study medication at the baseline visit (Visit 2, open label) and instructed to take 1 x 0.1 mg tablet each evening (Day 1) at bedtime until the next visit. Subjects who required an increase in total dose to 0.2 mg/day took 1 x 0.1 mg tablet (0.1 mg) in the morning and at bedtime until the next visit. Those who required a further increase in dose to 0.3 mg/day took 1 x 0.1 mg tablet in the morning and 2 x 0.1 mg tablets at bedtime until the next visit. Patient increasing dose to 0.4 mg/day were instructed to take 2 x 0.1 mg tablets in the morning and at bedtime until the next visit.
  Of 68 Subjects randomized to KAPVAY:
  24 (35.3%) oral dose of 0.4 mg/day 25 (36.8%) oral dose of 0.3 mg/day 14 (20.6%) oral dose of 0.2 mg/day 5 (7.4%) oral dose of 0.1 mg/day
- Subjects on Placebo: Subjects randomized to the placebo arm were tapered off their optimal dose of KAPVAY (as determined after a 4-week, open-label, dose optimization period) at weekly intervals in decrements of 0.1 mg/day until reaching the dose of 0 mg/day, and then received only placebo for the rest of the study
  Of 67 Subjects randomized to Placebo:
  26 (38.8%) oral dose of 0.4 mg/day 24 (35.8%) oral dose of 0.3 mg/day 15 (22.4%) oral dose of 0.2 mg/day 2 (3.0%) oral dose of 0.1 mg/day
Period: Overall Study
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Started | 68 | 67
Completed | 37 | 25
Not Completed | 31 | 42
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 5 | 21
Not completed — Protocol Violation | 6 | 4
Not completed — Lost to Follow-up | 6 | 3
Not completed — Other-Use of prohibited treatment | 0 | 2
Not completed — Other-Miscellaneous | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Subjects on KAPVAY (Clonidine Hydrochloride): Subjects in the KAPVAY arm received their optimal dose of KAPVAY (as determined after a 4-week, open-label, dose optimization period) for the duration of the 26-week randomized-withdrawal period
- Subjects on Placebo: Subjects randomized to the placebo arm were tapered off their optimal dose of KAPVAY (as determined after a 4-week, open-label, dose optimization period) at weekly intervals in decrements of 0.1 mg/day until reaching the dose of 0 mg/day, and then received only placebo for the rest of the study
- Total: Total of all reporting groups
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo | Total
Number analyzed (Participants) | 68 | 67 | 135
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.7 (2.77) | 10.9 (2.98) | 10.8 (2.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 43 | 51 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 20 | 32
  Not Hispanic or Latino | 56 | 47 | 103
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 14 | 37
  White | 37 | 50 | 87
  More than one race | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 40.49 (15.721) | 41.61 (16.978) | 41.05 (16.350)
Height [Mean (Standard Deviation); unit: cm] | 145.64 (17.737) | 145.45 (17.928) | 145.55 (17.833)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 18.29 (2.921) | 18.79 (3.485) | 18.54 (3.203)

OUTCOME MEASURES:

1. Primary Outcome: Long-term Maintenance of Efficacy of KAPVAY in Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD) as Measured by the Percentage of Treatment Failures in the KAPVAY vs. Placebo Groups
Description: Treatment failure a ≥30 percentage increase (worsening)(ADHD-RS-IV, clinician version) total score and a ≥2 point increase (worsening) in Clinical Global Impressions-Severity of Illness Scale (CGI-S) at any two consecutive visits during the randomized-withdrawal period.
  The ADHD-RS-IV of 2 subscales: inattention - 9 items and hyperactivity-impulsivity - 9 items. Each gives a score ranging from 0 (none, never or rarely) to 3 (severe, very often), for a total score ranging from 0 to 54 (higher score worse).
  The CGI-S is a 7-point scale,1 (Normal, not at all ill) to 7 (extremely ill patients).The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
Time Frame: From randomization to end of the randomized-withdrawal period (26 weeks)
Population: Double-Blind Full Analysis Set. This set included all randomized subjects who took at least 1 dose of study medication during the double blind (randomized-withdrawal) phase
Measure: Number; unit: % of Participants
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
% of Participants | 31 | 42

2. Secondary Outcome: To Evaluate the Long-term Efficacy of KAPVAY in Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD) as Measured by the Time to Treatment Failure From the Start of Randomized-withdrawal Period
Description: Time to treatment failure was calculated as follows: Treatment failure (not premature termination) = visit date where the failure criteria was met - visit 9 date + 1; Treatment failure (premature termination) = termination date - visit 9 date + 1
Time Frame: Time From randomization to treatment failure (up to 26 weeks)
Population: Double-Blind Full Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
days | 212 [84 to NA] — NA implies the median or the one or both limits in the confidence interval could not be estimated. | 75 [36 to 154]

3. Secondary Outcome: Long-term Efficacy of KAPVAY in Children and Adolescents With ADHD as Measured by the Change From Randomization to the End of the Randomized-withdrawal Period on the ADHD-Rating Scale-4th Edition (ADHD-RS-IV)
Description: The ADHD-RS-IV (clinician version), has been widely used as a measure of efficacy in clinical trials of treatments in children and adolescents with ADHD. It is derived from the 18 inattentive and hyperactive/impulsive diagnostic criteria for ADHD from the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR). The clinician version of the ADHD-RS-IV has a large base of normative data and has demonstrated reliability and discriminant validity in children and adolescents. The ADHD-RS-IV of 2 subscales: inattention - 9 items and hyperactivity-impulsivity - 9 items. Each gives a score ranging from 0 (none, never or rarely) to 3 (severe, very often), for a total score ranging from 0 to 54 (higher score worse and a lower score more favourable). Two subscales are summed.
Time Frame: From randomization to end of the randomized-withdrawal period (26 weeks)
Population: Double-Blind Full Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
scores on a scale | 3.0 (10.75) | 7.0 (12.30)

4. Secondary Outcome: Long-term Efficacy of KAPVAY in Children and Adolescents With ADHD as Measured by the Change From Randomization to the End of the Randomized-withdrawal Period on the Clinical Global Impressions-Severity of Illness Scale (CGI-S)
Description: The CGI-S is a clinician rated instrument designed to assess the subject's current illness state. The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  This rating is based upon observed and reported symptoms, behavior, and function in the past seven days.
Time Frame: From randomization to end of the randomized-withdrawal period (26 weeks)
Population: Double-Blind Full Analysis Set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
scores on a scale | 0.4 (1.20) | 0.9 (1.28)

5. Secondary Outcome: Long-term Efficacy of KAPVAY in Children and Adolescents With ADHD as Measured by the Change From Randomization to the End of the Randomized-withdrawal Period on the Weiss Functional Impairment Rating Scale-Parent (WFIRS-P)
Description: The WFIRS-P is designed to assess the impact of child's behavior or emotional problems on 7 domains related to function: Family (10 items), School Learning (4 items), School Behavior (6 items), Life Skills (10 items), Child's Self-concept (3 items), Social Activities (7 items), and Risky Activities (10 items). Each item was scored on a scale ranging from 0 ("never" or "not at all") to 3 ("very often" or "very much"). Each scale score was calculated as the average for that scale. The total score is the average of all non-missing items. Higher scores are associated with greater impact of disease on functioning.
Time Frame: From randomization to end of the randomized-withdrawal period (26 weeks)
Population: Double-Blind Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
units on a scale | 0.0 (0.34) | 0.0 (0.38)

6. Secondary Outcome: Long-term Efficacy of KAPVAY in Children and Adolescents With ADHD as Measured by the Change From Randomization to the End of the Randomized-withdrawal Period on the Epworth Sleepiness Scale for Children (ESS-C)
Description: Change in the ESS-C scale from randomization to end of randomized-withdrawal period. The ESS-C is a simple eight-tem Likert scale designed to assess daytime sleepiness in children aged 2-18 years. The scale takes less than two minutes to be completed by patient or by parent rating. Sleepiness is a common symptom in both medicated and unmedicated children with ADHD given the predominance of impaired sleep quality. The total score achieved when the chance of dozing in each situation is added up serves as the outcome measure.
  The ESS-C comprises 8 items describing various daytime activities. Item scores ranging from 0 ("would never doze or sleep") to 3 ("high chance of dozing or sleeping"). A total score is derived as the sum of the items, with higher total scores indicative of a greater level of sleepiness (worse outcome). Total scores range from 0 to 24.
Time Frame: From randomization to end of the randomized-withdrawal period (26 weeks)
Population: Double-Blind Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
units on a scale | -0.6 (3.18) | -0.6 (4.09)

7. Secondary Outcome: Long-term Safety of KAPVAY in Children and Adolescents With ADHD Based on the Assessment of Adverse Events (AEs), Serious Adverse Events (SAEs), AEs Leading to Study Drug Discontinuation, Clinically Significant Changes or Abnormalities in Vital Signs
Time Frame: From study start to study end (40 weeks)
Population: Double-Blind Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
Participants
  No. Subjects with At Least 1 Treatment-Emergent AE | 34 | 31
  Any Severe Treatment-Emergent AE (TEAE) | 2 | 0
  Any SAE | 0 | 2
  Treatment Emergent AE leading to discontinuation | 2 | 0
  Any Treatment-Related AE | 18 | 12
  Vital Signs Abnormalities | 3 | 1

8. Secondary Outcome: Long-term Safety of KAPVAY in Children and Adolescents With ADHD Based on the Assessment of Changes in the Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The outcome reported is the number of subjects that responded "Yes" to the question "Do you have a wish to be dead" at Visit 20.
  C-SSRS is a clinician-rated instrument designed to provide consistent and systematic assessment of both suicidal ideation and behavior within a study, as well as across studies. The scale is a feasible, low burden series of questions that appropriately assess and track all suicidal events, including ideation. Suicidal ideation is assessed according to yes/no responses to 5 questions of increasing severity (from a wish to die to an active thought of killing oneself with plan and intent) as follows:
  1. Wish to be Dead
  2. Non-Specific Active Suicidal Thoughts
  3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act
  4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan
  5. Active Suicidal Ideation with Specific Plan and Intent
Time Frame: Visit 20 (Week 40)
Population: Double-Blind Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Number analyzed (Participants) | 68 | 67
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Throughout the study
Arm/Group | Subjects on KAPVAY (Clonidine Hydrochloride) | Subjects on Placebo
Serious Adverse Events (participants affected / at risk) | 0/68 | 2/67
Other Adverse Events (participants affected / at risk) | 15/68 | 7/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on KAPVAY (Clonidine Hydrochloride) (N=68) | Subjects on Placebo (N=67)
Suicidal ideation (Psychiatric disorders) | 0 | 1
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects on KAPVAY (Clonidine Hydrochloride) (N=68) | Subjects on Placebo (N=67)
Somnolence (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 2 | 3
Sedation (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Electrocardiogram QT (Investigations) | 2 | 0
Weight increased (Investigations) | 2 | 0
Affect lability (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.